CLINICAL TRIAL: NCT07328555
Title: Site Randomized Clinical Trial of the Effect of Digital Otoscopy Versus Standard Otoscopy on the Diagnosis and Treatment of Otitis Media in Young Children
Brief Title: Digital Otoscopy Versus Standard Otoscopy on the Diagnosis and Treatment of Otitis Media in Young Children
Acronym: Wispr 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jon Hatoun, Director of Data Analytics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PPOC_Wispr 2
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Otitis Media; Antimicrobial Stewardship
Keywords: Otoscopy
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Intervention Model Description: Four enrolled practices:
  * Two will receive the intervention (digital otoscopy)
  * Two will not receive an intervention (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental: Digital Otoscopy (Experimental): Use of the Wispr digital otoscope to diagnose otitis media in place of a traditional visual otoscope
  Interventions: Device: Device: Digital Otoscope
- No intervention: Control (No Intervention): No intervention - standard otoscopy to be used

INTERVENTIONS:
Device: Device: Digital Otoscope — Use of the Wispr digital otoscope to diagnose otitis media in place of a standard visual otoscope
  Arms: Experimental: Digital Otoscopy

SUMMARY:
Randomized controlled trial involving 4 pediatric primary care practices in Massachusetts. Practices will be stratified by their OM diagnosis and treatment rate, with two practices randomly assigned to the intervention arm and two to the control arm.

For practices randomized to the intervention arm, their offices will be equipped with digital otoscopes (Wispr Digital Otoscope, WiscMed) in each exam room in place of traditional otoscopes. Clinicians in intervention practices will attend a two-hour initial training session on the use of digital otoscopy followed by two one-hour follow-up sessions held over a two-month run-in period prior to the study start to review best practices and troubleshoot any difficulties adapting to the new technology.

Upon completion of the run-in training period, a six-month data collection period will begin. The primary outcome will consist of a difference-in-difference analysis comparing the difference in the OM Treatment Index (OMTI) from the baseline period (October 1 through March 31, 2025) to the intervention period (October 1 through March 31, 2026) between the intervention practices and the control practices. The OMTI is a measure of the rate of diagnosis and antibiotic treatment of OM, specifically calculated as the number of cases with an OM diagnosis and systemic antibiotic prescribed divided by the number of visits with a diagnosis of any acute respiratory tract illness.

Secondary outcomes include analogous difference-in-difference comparisons of: 1) overall antibiotic courses prescribed; 2) overall days of antibiotics prescribed; and 3) a balancing measure of the rate of return visits with any acute respiratory tract illness diagnosis within 7 days of an index visit. Additionally, clinicians will be surveyed to assess confidence and satisfaction in diagnosing OM and preference for digital versus traditional otoscopy.

To incentivize participation, practices randomized to the control arm will be loaned digital otoscopes to use for six months at the conclusion of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. PPOC practices with 4-9 patient exam rooms, willing to commit to using digital otoscopy for 6 months.
2. Not currently using digital otoscopy.
3. Not involved in the network's previous digital otoscopy study

Exclusion Criteria:

* Currently using any digital otoscope

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in OMTI | 6 months
  Difference-in-differences analysis of the change in OMTI from baseline to the intervention period comparing the intervention arm to the control arm using logistic regression with nested random effect at the practice level.

SECONDARY OUTCOMES:
Change in overall antibiotic courses prescribed | 6 months
  Difference-in-differences analysis of the change in the overall number of antibiotic courses prescribed per 100 encounters (excluding well visits) comparing the intervention arm to the control arm, using logistic regression with nested random effect at the practice level.
Change in overall prescribed antibiotic days | 6 months
  Difference-in-differences analysis of the change in the overall number of prescribed antibiotic days per 100 encounters (excluding well visits) comparing the intervention arm to the control arm, using logistic regression with nested random effect at the practice level.
Return acute respiratory tract illness visits | Comparison between intervention and control arm of the proportion of patients with an index visit with an acute respiratory tract illness diagnosis who return to the PCP for a visit with an acute respiratory tract illness diagnosis within 7 days of index

CONTACTS AND LOCATIONS:
Overall Officials: Louis Vernacchio, MD, MSc, Study Director — Boston Children's Hospital
Locations (1):
- Pediatric Physicians' Organization at Children's, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Electronic health record data use for the study are property of the individual practices and may not be shard publicly without their expressed permission.